CLINICAL TRIAL: NCT04332302
Title: Effects of an Exercise Program on Physical Functionality and Frailty in Type 2 Diabetic Older Adults. Role of Circulating Concentration of PDEF and Differential Genes
Brief Title: Power Strength Training in Type 2 Diabetic Mellitus Older Adults
Acronym: DIAPOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Madrid (Other)
Collaborators: Spanish Society of Diabetes (Unknown); University of Castilla-La Mancha (Other); Castilla-La Mancha Health Service (Other)
Responsible Party: Principal Investigator, Amelia Guadalupe Grau, Principal Investigator, Technical University of Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SE1911600154
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Frailty
Keywords: Resistance Training; Quality of Life; Molecular Genetics; Skeletal Muscle
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power training group (Experimental): Participants will be enrolled in a resistance training program.
  Interventions: Other: Power resistance training
- Control group (No Intervention): Participants will be doing their normal life.

INTERVENTIONS:
Other: Power resistance training — Participants will take part in an intervention of 12 weeks duration in which they will train with musculation machines.
  Arms: Power training group

SUMMARY:
Diabetes is a disease with a high impact in the population older than 65 years old. Some indications suggest that diabetes in the old age aggravate the negative effects of ageing, as the loss of muscle mass and strength, bringing the patients to a situation of vulnerability and elevated risk of disability and death known as "frailty syndrome". Recently, scientists have observed that if older population train with musculation machines emphasising the muscular power, it is possible to have an impact on a disminution of frailty and restoring the physical functionality. This project deeps in the physiological and molecular mechanisms that underlie to improvements in the frail diabetic patients.

DETAILED DESCRIPTION:
It is hypothesised that:

1. High intensity training (strength-power) prescribed properly in an individualised form and supervised could influence significantly on the phenotypic response in the DM type 2: decreasing the level of clinical severity, disability and frailty, improving quality of life and glycaemic control, functional capacity and body composition (especially the muscle mass) of the diabetic patients (type 2) older than 65 years old.
2. Part of the training adaptations in diabetic patients (type 2) older than 65 years old could due to physiological conditions as the systemic level of biomarkers as PDEF in these patients.
3. Part of the training adaptations in diabetic patients (type 2) could be influenced by the characterisation of associated genes to the different types of DM type 2 recently characterised.

The principal aims are:

1. To evaluate the effectiveness of a novel intervention based on strength-power exercise in individuals older than 65 years old with DM type 2 and frailty in term of: level of clinical severity, disability, glycaemic control, quality of life, functional capacity, state of frailty and body composition.
2. To establish whether PDEF serves as diagnostic and prediction biomarker to training response, providing an objective and accessible method that would stratify the response to the intervention helping with the patients screening.
3. To determine the role of characterised genetic variants in the different subgroups of DM type 2 in the level of response to the training stimuli.

Study design Longitudinal intervention stratified study, controlled and single-blinded, with a group of intervention and control group.

Based on data from a previous study recently published by the collaborators of this project. The sample size was calculated to get statistically significant differences in the physical functionality using ANCOVA and performing a bilateral contrast with alpha=0.05 of the effect of the group (with any of the independent variables), and it is needed 30 subjects by group (total n=60) to get a statistical power of 80%, with a partial eta ≥ 0.101 (value that corresponds with the size of the moderate effect).

Exercise program The intervention period will have a duration of 12 weeks, in which the training group will perform 2 sessions per week (24 sessions in total), while the control group will not perform any type of intervention, following their normal lifes and the habitual medical cares. The experimental group will perform a program focused on the muscle power training, in which there will be included exercise of upper limbs (chest press) and lower limbs (leg press). The exercises will be performed in muscle-building machines available in the reference institutions of the collaborators. It is important to point out that the intensity in the exercises will be individualised for any patient through a test of determination of muscle power validated previously by the consortium of researchers and the subjects will perform the exercises at this intensity at which the subjects will develop their maximal muscle performance, with the performance of 3-4 bouts of 8 repetitions in each exercise. After the third week of intervention, it will be put the attention to the speed of execution. The duration of each session has been estimated in 20-30 minutes.

Finally, the subjects in the control group will serve to compare the interventions with exercise and the clinical conventional treatment, as well as to determine whether the training program is able to restore the functional capacity in a similar way in diabetic patients without frailty.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent.
* Older than 65 years old with Type 2 Diabetes Mellitus diagnosed in a minimum of 2 previous years.
* Being diagnosed frail, pre-frail or no frail.

Exclusion Criteria:

* Barthel's index lower than 60 points.
* Incapacity to complete the SPPB fitness test.
* Score lower than 20 points in the Mini Mental State Examination.
* Cardiovascular event in the previous 6 months following the New York Heart Association (NYHA) classification.
* Patients clinically unstable by the investigator's judgement.
* Terminal disease (life expectancy lower than 6 months).
* Participation in another study that could interfere in the results of the current research.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Glycosylated Hemoglobin (Hemoglobin A1c) at 12 weeks | 0 and 12 weeks.
  Percentage
Change from Baseline Homeostasis Model Assessment - Beta cells (HOMA2-B) at 12 weeks | 0 and 12 weeks.
  Percentage
Change from Baseline Homeostasis Model Assessment - Insuline Resistance (HOMA2-IR) at 12 weeks | 0 and 12 weeks.
  Percentage
Change from Baseline Fried frailty score at 6 and 12 weeks | 0, 6 and 12 weeks.
  Level of frailty assessed by Fried Criteria. Intermediate or prefrail: 1 or 2 criteria present. Positive for frailty phenotype: ≥3 criteria present.
Change from Baseline Functional capacity at 6 and 12 weeks | 0, 6 and 12 weeks.
  Level of functional capacity assessed by the test SPPB. Scores 0-3: Very low physical function; Scores 4-6: Low physical function; Scores 7-9: Moderate physical function; Scores 10-12: High physical function
Change from Baseline Disability at 6 and 12 weeks | 0, 6 and 12 weeks.
  Level of disability assessed by the Barthel test. A participant scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities.
Functional mobility at 6 and 12 weeks | 0, 6 and 12 weeks.
  Level of functional mobility assessed by the Lawton test. A scale from 0 to 8, expressing higher scores better levels of independence.
Change from Baseline Muscular power at 6 and 12 weeks | 0, 6 and 12 weeks.
  Watts.
Change from Baseline Levels of strength at 6 and 12 weeks | 0, 6 and 12 weeks.
  Load (kg).
Change from Baseline Bone Mineral Density at 12 weeks | 0 and 12 weeks.
  g/cm3
Change from Baseline Pigment Epitelium Derived Factor (PEDF) at 12 weeks | 0 and 12 weeks.
  Circulating level of PDEF assessed by Western Blot.
Genotyping of TCF7L2 (rs7903146) | 0 week.
  Assessed by Real-time PCR.
Genotyping of TM6SF2 (rs10401969) | 0 week.
  Assessed by Real-time PCR.
Genotyping of HLA (rs2854275) | 0 week.
  Assessed by Real-time PCR.

SECONDARY OUTCOMES:
Change from Baseline Body Mass Index at 6 and 12 weeks | 0, 6 and 12 weeks.
  Kg by square meters.
Change from Baseline Waist circumference at 6 and 12 weeks | 0, 6 and 12 weeks.
  Meters.
Change from Baseline Blood pressure (systolic and diastolic) at 6 and 12 weeks | 0, 6 and 12 weeks.
  mmHg.
Change from Baseline Concentration of Triglycerides at 12 weeks | 0 and 12 weeks.
  mg/dL.
Change from Baseline Concentration of Total Cholesterol at 12 weeks | 0 and 12 weeks.
  mg/dL.
Change from Baseline Concentration of HDL Cholesterol at 12 weeks | 0 and 12 weeks.
  mg/dL.
Change from Baseline Concentration of LDL Cholesterol at 12 weeks | 0 and 12 weeks.
  mg/dL.
Change from Baseline Subjective level of quality of life at 12 weeks | 0 and 12 weeks.
  Level of quality of life assessed by the test EuroQoL index, EQ-5D-5L. The score is the time trade-off (TTO). Scale from 11111 to 55555 being the higher the best health related quality of life.
Change from Baseline Physical activity at 12 weeks | 0 and 12 weeks.
  Accelerometry, counts/min.
Change from Baseline Balance at 12 weeks | 0 and 12 weeks.
  Level of balance assessed in a force platform. Newtons.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Guadalupe Grau, PhD, Principal Investigator — Technical University of Madrid; Carmen Ramírez Castillejo, PhD, Study Chair — Technical University of Madrid; Marcela González Gross, Professor, Study Director — Technical University of Madrid
Locations (1):
- Instituto Nacional de Educación Física, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individualised report to all the participants after the completion of the study.
Supporting Information: Analytic Code
Time Frame: At the end of the intervention.
Access Criteria: The participants who have accepted to have the report.

REFERENCES:
- [Background] Guadalupe-Grau A, Carnicero JA, Gomez-Cabello A, Gutierrez Avila G, Humanes S, Alegre LM, Castro M, Rodriguez-Manas L, Garcia-Garcia FJ. Association of regional muscle strength with mortality and hospitalisation in older people. Age Ageing. 2015 Sep;44(5):790-5. doi: 10.1093/ageing/afv080. Epub 2015 Jul 11. PMID 26163682
- [Background] Garcia-Garcia FJ, Carcaillon L, Fernandez-Tresguerres J, Alfaro A, Larrion JL, Castillo C, Rodriguez-Manas L. A new operational definition of frailty: the Frailty Trait Scale. J Am Med Dir Assoc. 2014 May;15(5):371.e7-371.e13. doi: 10.1016/j.jamda.2014.01.004. Epub 2014 Mar 2. PMID 24598478
- [Background] Garcia-Garcia FJ, Gutierrez Avila G, Alfaro-Acha A, Amor Andres MS, De Los Angeles De La Torre Lanza M, Escribano Aparicio MV, Humanes Aparicio S, Larrion Zugasti JL, Gomez-Serranillo Reus M, Rodriguez-Artalejo F, Rodriguez-Manas L; Toledo Study Group. The prevalence of frailty syndrome in an older population from Spain. The Toledo Study for Healthy Aging. J Nutr Health Aging. 2011 Dec;15(10):852-6. doi: 10.1007/s12603-011-0075-8. PMID 22159772
- [Background] Losa-Reyna J, Baltasar-Fernandez I, Alcazar J, Navarro-Cruz R, Garcia-Garcia FJ, Alegre LM, Alfaro-Acha A. Effect of a short multicomponent exercise intervention focused on muscle power in frail and pre frail elderly: A pilot trial. Exp Gerontol. 2019 Jan;115:114-121. doi: 10.1016/j.exger.2018.11.022. Epub 2018 Dec 4. PMID 30528641
- [Background] Alcazar J, Rodriguez-Lopez C, Ara I, Alfaro-Acha A, Rodriguez-Gomez I, Navarro-Cruz R, Losa-Reyna J, Garcia-Garcia FJ, Alegre LM. Force-velocity profiling in older adults: An adequate tool for the management of functional trajectories with aging. Exp Gerontol. 2018 Jul 15;108:1-6. doi: 10.1016/j.exger.2018.03.015. Epub 2018 Mar 20. PMID 29567100
- [Background] Alcazar J, Guadalupe-Grau A, Garcia-Garcia FJ, Ara I, Alegre LM. Skeletal Muscle Power Measurement in Older People: A Systematic Review of Testing Protocols and Adverse Events. J Gerontol A Biol Sci Med Sci. 2018 Jun 14;73(7):914-924. doi: 10.1093/gerona/glx216. PMID 29309534
- [Background] Alcazar J, Rodriguez-Lopez C, Ara I, Alfaro-Acha A, Manas-Bote A, Guadalupe-Grau A, Garcia-Garcia FJ, Alegre LM. The Force-Velocity Relationship in Older People: Reliability and Validity of a Systematic Procedure. Int J Sports Med. 2017 Dec;38(14):1097-1104. doi: 10.1055/s-0043-119880. Epub 2017 Nov 10. PMID 29126339
- [Background] Guadalupe-Grau A, Aznar-Lain S, Manas A, Castellanos J, Alcazar J, Ara I, Mata E, Daimiel R, Garcia-Garcia FJ. Short- and Long-Term Effects of Concurrent Strength and HIIT Training in Octogenarians with COPD. J Aging Phys Act. 2017 Jan;25(1):105-115. doi: 10.1123/japa.2015-0307. Epub 2016 Aug 24. PMID 27402660

DOCUMENTS (1):
  • Informed Consent Form (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT04332302/ICF_000.pdf